CLINICAL TRIAL: NCT07131293
Title: European Registry Study on Lymphatic Interventions: Towards Standardized Care in CHD-Related Lymphatic Disorders
Brief Title: European Registry Study on Lymphatic Interventions
Acronym: EURO-LYMPH
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: UZ Leuven, Leuven, Belgium (Unknown); UCL Bruxelles (Unknown); Lund University Hospital (Other); University Hospital Schleswig-Holstein (Other); University Hospital, Aachen (Other); Deutsches Herzzentrum Muenchen (Other); Universitätsklinikum Erlangen, Erlangen, Bayern, Germany (Unknown); UZ Gent, Belgium (Unknown); Hospital for Children and Adolescents, University of Helsinki (Unknown); Hospital Universitari Vall d'hebron Barcelona, Spain (Unknown); Children's University Hospital, Ireland (Other); Evelina London Children's Hospital (Unknown); Guy's and St Thomas' NHS Foundation Trust (Other); Bambin Gesù Hospital IRCCS, Rome, Italy (Unknown)
Responsible Party: Principal Investigator, Sanam Safi-Rasmussen, Sanam Safi-Rasmussen, MD & PhD-fellow, Rigshospitalet, Denmark
Other Study IDs: R-25051744
Record Dates: First submitted 2025-07-29; First posted 2025-08-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Lymphatic Disorders; Plastic Bronchitis; Protein Losing Enteropathy; Chylothorax; Lymphatic Abnormalities
Keywords: Lymphatic complications; Multicenter study; Plastic bronchitis; Protein Losing Enteropathy; Chylothorax
MeSH Terms: conditions — Lymphatic Diseases; Protein-Losing Enteropathies; Chylothorax; Lymphatic Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lymph intervention
  Interventions: Procedure: Lymphatic intervention

INTERVENTIONS:
Procedure: Lymphatic intervention — This intervention was made as part of their clinical treatment.

SUMMARY:
This European multicenter observational study aims to evaluate the real-world use, timing, and outcomes of lymphatic interventions in patients with congenital heart disease and/or primary lymphatic disorders. The study will examine the effectiveness of diagnostic imaging and interventional techniques, such as lymphatic embolization, in improving clinical symptoms, biomarkers, and fluid-related complications. The central question is whether early diagnosis and targeted intervention can lead to clinically meaningful improvements and reduced need for reintervention. Data collected retrospectively and prospectively from participating centers will help identify predictors of outcome, assess disease severity, and inform standardized diagnostic and therapeutic pathways across Europe.

DETAILED DESCRIPTION:
This is a prospective, multicenter observational study with retrospective components. The study population includes patients who have undergone or are undergoing lymphatic imaging diagnostics and lymphatic interventions at participating centers across Europe. Patients are included both retrospectively (from medical records) and prospectively as part of their routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age with a confirmed central lymphatic disorder, either in the context of CHD or as a primary lymphatic disorder, verified through lymphatic diagnostics (e.g. lymphatic imaging or relevant biomarkers).
* Patients who have undergone, or are undergoing, diagnostic lymphatic imaging and/or interventional procedures for their lymphatic disorder.
* Patients who are receiving, or have received, conservative (non-interventional) management for their lymphatic disorder.

Exclusion Criteria:

* Patients with isolated peripheral lymphatic disorders not involving the central lymphatic system.
* Patients with acute postoperative iatrogenic chylothorax (<3-4 weeks duration and not requiring intervention).
* Patients without sufficient clinical documentation to confirm diagnosis, treatment, or follow-up.
* Patients who decline, or whose legal guardians decline, to provide informed consent (for prospective inclusion).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be identified from pediatric and adult congenital cardiology and lymphatic referral centers across Europe. The study population includes patients of any age with congenital heart disease (CHD) and associated central lymphatic complications (such as plastic bronchitis, protein-losing enteropathy, or chylothorax), as well as patients with primary central lymphatic disorders. Patients are included from tertiary care institutions that perform lymphatic imaging and/or interventions and will be enrolled retrospectively from existing clinical records and prospectively during routine care.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Change in Symptoms Following Lymphatic Intervention, assessed by: | From time of treatment to yearly follow-up up to 5 years.
  Patient-reported or physician-assessed symptoms (e.g., cough, diarrhea, dyspnea) will be categorized as normalized, improved, unchanged, or worsened compared to baseline.
  Unit of Measure:
  Symptom status category (normalized / improved / unchanged / worsened)
Change in Objective Biomarkers Following Lymphatic Intervention | From time of treatment to yearly follow-up up to 5 years.
  Objective clinical findings (e.g., serum albumin level, lymphocyte count, fluid accumulation) will be categorized as normalized, improved, unchanged, or worsened compared to baseline.
  Unit of Measure:
  Biomarker status category (normalized / improved / unchanged / worsened)
Composite improvement: | From time of treatment to yearly follow-up up to 5 years.
  ≥50% reduction in presenting symptoms and/or ≥20% improvement in key biomarkers (e.g., serum albumin, lymphocyte count etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke E Hjortdal, Professor, Study Director — Rigshospitalet, Denmark; Michael Rahbek Schmidt, Ass. professor, PhD, DMSc, Study Director — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No